CLINICAL TRIAL: NCT03385486
Title: A Phase 1 Multi-Center Dose-Escalation Study of the Safety, Tolerability and Early Efficacy of TBX-3400 in Patients With Stage III and IV Melanoma Resistant or Refractory to Immune Checkpoint Inhibitors
Brief Title: Study of TBX-3400 in Patients With Stage III and IV Melanoma Resistant or Refractory to Immune Checkpoint Inhibitors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiga Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TBX-3400-001
Record Dates: First submitted 2017-12-03; First posted 2017-12-28 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Stage III Melanoma; Stage IV Melanoma
Keywords: Melanoma; Resistant; Refractory
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: The study will consist of a Dose Escalation Phase and a Dose Expansion Phase. TBX-3400 will be administered on Day 1 of each treatment cycle and can be repeated.
  In the Dose Escalation Phase, a "3+3" design will be employed. Each dose cohort will initially enroll 3 patients. Enrollment and treatment of the first 3 patients in the first cohort will be staggered to allow for evaluation of safety. After each cohort has been enrolled and all patients in the cohort have completed Cycle 1, a Data Safety Monitoring Committee will review cumulative safety data to determine whether to proceed with further dose escalation.
  Each cohort may be expanded in groups of 3 patients to a maximum of 12 patients. Up to six TBX 3400 dose levels will be evaluated during the Dose Escalation Phase of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TBX-3400 (Experimental): TBX-3400 by intravenous infusion
  Interventions: Biological: TBX-3400

INTERVENTIONS:
Biological: TBX-3400 — Autologous transfusion

SUMMARY:
This is a study of transfusion of TBX-3400 in patients with stage III and IV melanoma resistant or refractory to Immune Checkpoint Inhibitors.

The patient's own blood cells are exposed to a protein that has been shown in the laboratory to result in anti-tumor activity.

The study hypothesis is that TBX-3400 cells will enhance anti-tumor activity and improve the body's immune response.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in the study:

1. Histopathologically confirmed diagnosis of advanced, unresectable or metastatic malignant melanoma
2. Male or female patients age 18 or older
3. Previously treated with checkpoint inhibitor therapy either alone or in combination with either stable disease or progressive disease per RECIST version 1.1 (there is no minimum treatment duration for patients who have progressive disease while on checkpoint inhibitor therapy)
4. Measurable or evaluable disease by RECIST version 1.1
5. Capable of understanding and complying with protocol requirements
6. A life expectancy of greater than 24 weeks at Screening
7. ECOG Performance Status of 0 to 2
8. Written informed consent from the patient or the patient's legally acceptable representative prior to the initiation of any study procedures
9. Adequate bone marrow, liver, and renal function as defined below:

   * hemoglobin ≥8.0 g/dL (transfusions allowed)
   * absolute neutrophil count ≥1500/µL
   * platelet count ≥100,000/µL (transfusions allowed)
   * alanine transaminase and aspartate transaminase ≤3.0 times the upper limit of normal (ULN), or ≤5 times ULN for patients with known hepatic metastases
   * total serum bilirubin ≤1.5 x the ULN; ≤2.0 x the ULN if liver metastases are present; patients with a known history of Gilbert's syndrome (≤3.0 x the ULN) and/or isolated elevations of indirect bilirubin are eligible for study participation
   * estimated glomerular filtration rate ≥50 mL/min/1.73 m^2 (using Cockcroft Gault formula)

Exclusion Criteria:

Patients who meet any of the following criteria will not be eligible for participation in the study:

1. Pregnant or breast feeding
2. Developed immune-related toxicity while on prior checkpoint inhibitor therapy that has not yet returned to Grade 1 or better
3. Require systemic pharmacologic doses of corticosteroids at or above the equivalent of 10 mg/day of prednisone; replacement doses, topical, ophthalmologic and inhalational steroids are permitted
4. Active, symptomatic central nervous system (CNS) metastases. Patients with CNS metastases are eligible for the trial if the metastases have been treated by surgery and/or radiotherapy and the patient is off corticosteroids and is neurologically stable for at least 7 days prior to screening
5. Any concurrent uncontrolled illness, including mental illness or substance abuse which in the opinion of the investigator would make the patient unable to cooperate or participate in the trial
6. Severe uncontrolled cardiac disease within 3 months of study entry, including unstable or new onset angina, myocardial infarction or cerebrovascular accident
7. Women of childbearing potential who are unable or unwilling to use an acceptable method of contraception
8. Known infection with human immunodeficiency virus (HIV) that is not well controlled on anti-retroviral therapy as defined by HIV RNA more than 400 copies/mL or severely symptomatic
9. Presence of Hepatitis B and/or Hepatitis C active infection
10. Symptomatic congestive heart failure, defined as New York Heart Association Class II or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-06-02 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs), including the incidence of dose-limiting toxicities (DLTs), graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | 26 months
  Adverse events from subject reporting

SECONDARY OUTCOMES:
Tumor responses as defined by RECIST version 1.1 | 26 months
  Tumor measurements to assess disease state
Tumor responses as defined by irRECIST | 26 months
  Tumor measurements to assess disease state
Assessment of concentrations of certain chemokines, such as cluster of differentiation 69 (CD69), as biomarkers of activity of TBX-3400 | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Presence and/or concentration of anti TBX-3400 antibodies | 26 months
  Measure of immunogenicity of TBX-3400

OTHER OUTCOMES:
Quantification of the concentration of interleukin-1 (IL-1) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interleukin-6 (IL-6) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon-alpha (INF-α) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon gamma inducible protein 10 kD (IP-10) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of interferon-gamma (IFN-γ) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400
Quantification of the concentration of transforming growth factor-beta (TGF-ß) in plasma | 26 months
  Preliminary efficacy assessment to measure activity of TBX-3400

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No